CLINICAL TRIAL: NCT02246101
Title: Renal and Cardiovascular Impairment in WTC Responders: Implications for Diagnosis and Treatment
Brief Title: World Trade Center (WTC) RENAL
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GCO 13-1847; 1U01OH010716-01 (NIH)
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Disease; Cardiopulmonary Disease; Renal Disease; Cardiovascular Disease
Keywords: cardiac disease; cardiopulmonary disease; renal disease; albuminuria; cardiovascular disease; CVD; particulate matter
MeSH Terms: conditions — Heart Diseases; Pulmonary Heart Disease; Kidney Diseases; Cardiovascular Diseases; Albuminuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- WTC responders: WTC responders who were enrolled in the WTC-CHEST program.

SUMMARY:
Environmental toxins exert damaging health effects in workers. Thousands of responders who worked or volunteered on the World Trade Center (WTC) rescue and recovery effort following the September 11, 2001 attacks suffer from health conditions or may be at increased risk for worsening health. In a pilot study, investigators identified the first evidence of kidney damage in subjects with very high exposure at Ground Zero. Specifically, noted was a preliminary association between the intensity of particulate matter exposure and albuminuria, a marker of early chronic kidney disease (CKD), systemic endothelial dysfunction, and increased cardiovascular risk.

The long-term goal is to minimize the risk of CKD and cardiovascular disease (CVD) among individuals exposed to inhaled toxins. The primary objective of this research is to quantify the risk of kidney damage among first responders to the WTC attack and to determine the relationship to particulate matter exposure as well as determine an association between renal and cardiovascular damage in first responders and to explore potential mechanisms. The central hypothesis is that exposure to inhaled particulate matter causes systemic inflammation and endothelial dysfunction that result in chronic kidney and cardiovascular damage. This hypothesis will be investigated in a subgroup of participants from a previously conducted NIOSH-funded study "Pulmonary Function Abnormalities, Diastolic Dysfunction and WTC Exposure: Implications for Diagnosis and Treatment" ("WTC-CHEST," PI Mary Ann McLaughlin).

The proposed study will capitalize on unique resources in WTC-CHEST, including the standardized collection of data on particulate matter exposure and shared risk factors for CKD and cardiovascular disease, and cardiopulmonary function testing. The output from this proposal is anticipated to have a broad impact on understanding the health effects of inhaled particulate matter.

DETAILED DESCRIPTION:
Specific Aim 1. To quantify the risk of kidney damage and the relationship to particulate matter exposure among first responders to the WTC attack.

Urine samples will be collected on 2 occasions for albumin and creatinine. The investigators will define clinically relevant albuminuria as a UACR ≥30 mg/g. If, as hypothesized, the investigators find that albuminuria is more common among WTC responders, this simple and non-invasive measure may be useful in monitoring programs to identify responders at increased risk for adverse outcomes. eGFR will be calculated using the Chronic Kidney Disease Epidemiology Consortium (CKD-EPI) equations.

Specific Aim 2. To examine the relationship between kidney damage and cardiac structure and function among first responders to the WTC attack.

Cardiovascular Disease Risk Screening In order to identify an independent relationship between CKD and cardiac dysfunction, the investigators will comprehensively evaluate potential confounders. Participants will undergo an evaluation of traditional CVD risk factors as accounted for in both the Framingham Risk Score and Reynold's score (medical history, medication use and baseline risk for CVD: smoking status, family history of premature coronary disease, blood pressure, heart rate, height, weight, waist, hip and neck circumference). Laboratory evaluation will include: lipid panel, complete blood count, HbA1C, serum creatinine and cystatin C. Standard questionnaires on chest pain, shortness of breath, depression, sleep apnea and stress, IPSS.

Specific Aim 3. To explore potential mechanisms for kidney and cardiovascular damage among first responders to the WTC attack.

An established marker of systemic inflammation, serum hsCRP, will be measured in all participants. Flow-mediated dilatation, a validated non-invasive measure of endothelial function, will be measured in a subgroup of participants. Heavy metal assays will be performed and will be compared between participants with and without evidence of kidney damage (albuminuria or decreased eGFR) or proximal tubular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* WTC responders who were enrolled in the WTC-CHEST program.
* World Trade Center responders who are currently enrolled in the World Trade Center Health Program-Clinical Center of Excellence, formerly known as the WTC Medical Monitoring and Treatment Program
* Over the age of 39 years

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: World Trade Center rescue and recovery workers and volunteers who are enrolled in the World Trade Center Health Program-Clinical Center of Excellence, formerly known as the Medical Monitoring Treatment Program and were subsequently enrolled in the WTC-CHEST program.
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) | Day 1
  Kidney Function - To quantify the risk of kidney damage and the relationship to particulate matter exposure among first responders to the WTC attack.

SECONDARY OUTCOMES:
Echocardiography | Day 1
  Cardiac structure - To examine the relationship between kidney damage and cardiac structure and function among first responders to the WTC attack.
Urine Albumin level | Day 1
  Cardiac function - To examine the relationship between kidney damage and cardiac structure and function among first responders to the WTC attack.
High Sensitivity C-reactive Protein (hsCRP) | Day 1
  Endothelial Dysfunction - To explore potential mechanisms for kidney and cardiovascular damage among first responders to the WTC attack.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann McLaughlin, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Wisnivesky JP, Teitelbaum SL, Todd AC, Boffetta P, Crane M, Crowley L, de la Hoz RE, Dellenbaugh C, Harrison D, Herbert R, Kim H, Jeon Y, Kaplan J, Katz C, Levin S, Luft B, Markowitz S, Moline JM, Ozbay F, Pietrzak RH, Shapiro M, Sharma V, Skloot G, Southwick S, Stevenson LA, Udasin I, Wallenstein S, Landrigan PJ. Persistence of multiple illnesses in World Trade Center rescue and recovery workers: a cohort study. Lancet. 2011 Sep 3;378(9794):888-97. doi: 10.1016/S0140-6736(11)61180-X. PMID 21890053
- [Background] Landrigan PJ, Lioy PJ, Thurston G, Berkowitz G, Chen LC, Chillrud SN, Gavett SH, Georgopoulos PG, Geyh AS, Levin S, Perera F, Rappaport SM, Small C; NIEHS World Trade Center Working Group. Health and environmental consequences of the world trade center disaster. Environ Health Perspect. 2004 May;112(6):731-9. doi: 10.1289/ehp.6702. PMID 15121517
- [Background] Lioy PJ, Weisel CP, Millette JR, Eisenreich S, Vallero D, Offenberg J, Buckley B, Turpin B, Zhong M, Cohen MD, Prophete C, Yang I, Stiles R, Chee G, Johnson W, Porcja R, Alimokhtari S, Hale RC, Weschler C, Chen LC. Characterization of the dust/smoke aerosol that settled east of the World Trade Center (WTC) in lower Manhattan after the collapse of the WTC 11 September 2001. Environ Health Perspect. 2002 Jul;110(7):703-14. doi: 10.1289/ehp.02110703. PMID 12117648
- [Background] McGee JK, Chen LC, Cohen MD, Chee GR, Prophete CM, Haykal-Coates N, Wasson SJ, Conner TL, Costa DL, Gavett SH. Chemical analysis of World Trade Center fine particulate matter for use in toxicologic assessment. Environ Health Perspect. 2003 Jun;111(7):972-80. doi: 10.1289/ehp.5930. PMID 12782501
- [Background] Clarke RH, Holm LE. The Commission's policy on the environment. Ann ICRP. 2003;33(3):201-3. No abstract available. PMID 14582477
- [Background] Solan S, Wallenstein S, Shapiro M, Teitelbaum SL, Stevenson L, Kochman A, Kaplan J, Dellenbaugh C, Kahn A, Biro FN, Crane M, Crowley L, Gabrilove J, Gonsalves L, Harrison D, Herbert R, Luft B, Markowitz SB, Moline J, Niu X, Sacks H, Shukla G, Udasin I, Lucchini RG, Boffetta P, Landrigan PJ. Cancer incidence in world trade center rescue and recovery workers, 2001-2008. Environ Health Perspect. 2013 Jun;121(6):699-704. doi: 10.1289/ehp.1205894. Epub 2013 Apr 23. PMID 23613120
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Bash LD, Erlinger TP, Coresh J, Marsh-Manzi J, Folsom AR, Astor BC. Inflammation, hemostasis, and the risk of kidney function decline in the Atherosclerosis Risk in Communities (ARIC) Study. Am J Kidney Dis. 2009 Apr;53(4):596-605. doi: 10.1053/j.ajkd.2008.10.044. Epub 2008 Dec 24. PMID 19110358
- [Background] Gansevoort RT, Correa-Rotter R, Hemmelgarn BR, Jafar TH, Heerspink HJ, Mann JF, Matsushita K, Wen CP. Chronic kidney disease and cardiovascular risk: epidemiology, mechanisms, and prevention. Lancet. 2013 Jul 27;382(9889):339-52. doi: 10.1016/S0140-6736(13)60595-4. Epub 2013 May 31. PMID 23727170
- [Background] Peters A, von Klot S, Heier M, Trentinaglia I, Hormann A, Wichmann HE, Lowel H; Cooperative Health Research in the Region of Augsburg Study Group. Exposure to traffic and the onset of myocardial infarction. N Engl J Med. 2004 Oct 21;351(17):1721-30. doi: 10.1056/NEJMoa040203. PMID 15496621
- [Background] Pope CA 3rd, Burnett RT, Thurston GD, Thun MJ, Calle EE, Krewski D, Godleski JJ. Cardiovascular mortality and long-term exposure to particulate air pollution: epidemiological evidence of general pathophysiological pathways of disease. Circulation. 2004 Jan 6;109(1):71-7. doi: 10.1161/01.CIR.0000108927.80044.7F. Epub 2003 Dec 15. PMID 14676145
- [Background] Rossi G, Vigotti MA, Zanobetti A, Repetto F, Gianelle V, Schwartz J. Air pollution and cause-specific mortality in Milan, Italy, 1980-1989. Arch Environ Health. 1999 May-Jun;54(3):158-64. doi: 10.1080/00039899909602254. PMID 10444036
- [Background] Brook RD, Rajagopalan S, Pope CA 3rd, Brook JR, Bhatnagar A, Diez-Roux AV, Holguin F, Hong Y, Luepker RV, Mittleman MA, Peters A, Siscovick D, Smith SC Jr, Whitsel L, Kaufman JD; American Heart Association Council on Epidemiology and Prevention, Council on the Kidney in Cardiovascular Disease, and Council on Nutrition, Physical Activity and Metabolism. Particulate matter air pollution and cardiovascular disease: An update to the scientific statement from the American Heart Association. Circulation. 2010 Jun 1;121(21):2331-78. doi: 10.1161/CIR.0b013e3181dbece1. Epub 2010 May 10. PMID 20458016
- [Background] Hoffmann B, Moebus S, Mohlenkamp S, Stang A, Lehmann N, Dragano N, Schmermund A, Memmesheimer M, Mann K, Erbel R, Jockel KH; Heinz Nixdorf Recall Study Investigative Group. Residential exposure to traffic is associated with coronary atherosclerosis. Circulation. 2007 Jul 31;116(5):489-96. doi: 10.1161/CIRCULATIONAHA.107.693622. Epub 2007 Jul 16. PMID 17638927
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Gansevoort RT, Matsushita K, van der Velde M, Astor BC, Woodward M, Levey AS, de Jong PE, Coresh J; Chronic Kidney Disease Prognosis Consortium. Lower estimated GFR and higher albuminuria are associated with adverse kidney outcomes. A collaborative meta-analysis of general and high-risk population cohorts. Kidney Int. 2011 Jul;80(1):93-104. doi: 10.1038/ki.2010.531. Epub 2011 Feb 2. PMID 21289597
- [Background] Levy D, Garrison RJ, Savage DD, Kannel WB, Castelli WP. Left ventricular mass and incidence of coronary heart disease in an elderly cohort. The Framingham Heart Study. Ann Intern Med. 1989 Jan 15;110(2):101-7. doi: 10.7326/0003-4819-110-2-101. PMID 2521199
- [Background] Diamond JA, Phillips RA. Hypertensive heart disease. Hypertens Res. 2005 Mar;28(3):191-202. doi: 10.1291/hypres.28.191. PMID 16097361
- [Background] O'Neill MS, Diez-Roux AV, Auchincloss AH, Franklin TG, Jacobs DR Jr, Astor BC, Dvonch JT, Kaufman J. Airborne particulate matter exposure and urinary albumin excretion: the Multi-Ethnic Study of Atherosclerosis. Occup Environ Med. 2008 Aug;65(8):534-40. doi: 10.1136/oem.2007.035238. Epub 2007 Nov 21. PMID 18032533
- [Background] Kramer H, Jacobs DR Jr, Bild D, Post W, Saad MF, Detrano R, Tracy R, Cooper R, Liu K. Urine albumin excretion and subclinical cardiovascular disease. The Multi-Ethnic Study of Atherosclerosis. Hypertension. 2005 Jul;46(1):38-43. doi: 10.1161/01.HYP.0000171189.48911.18. Epub 2005 Jun 13. PMID 15956113
- [Background] Mani V, Wong SK, Sawit ST, Calcagno C, Maceda C, Ramachandran S, Fayad ZA, Moline J, McLaughlin MA. Relationship between particulate matter exposure and atherogenic profile in "Ground Zero" workers as shown by dynamic contrast enhanced MR imaging. Int J Cardiovasc Imaging. 2013 Apr;29(4):827-33. doi: 10.1007/s10554-012-0154-x. Epub 2012 Nov 23. PMID 23179748
- [Background] Ekong EB, Jaar BG, Weaver VM. Lead-related nephrotoxicity: a review of the epidemiologic evidence. Kidney Int. 2006 Dec;70(12):2074-84. doi: 10.1038/sj.ki.5001809. Epub 2006 Oct 25. PMID 17063179
- [Background] Jarup L, Hellstrom L, Alfven T, Carlsson MD, Grubb A, Persson B, Pettersson C, Spang G, Schutz A, Elinder CG. Low level exposure to cadmium and early kidney damage: the OSCAR study. Occup Environ Med. 2000 Oct;57(10):668-72. doi: 10.1136/oem.57.10.668. PMID 10984338
- [Background] Lin HH, Chou SA, Yang HY, Hwang YH, Kuo CH, Kao TW, Lo TC, Chen PC. Association of blood lead and mercury with estimated GFR in herbalists after the ban of herbs containing aristolochic acids in Taiwan. Occup Environ Med. 2013 Aug;70(8):545-51. doi: 10.1136/oemed-2012-101066. Epub 2013 May 23. PMID 23703822
- [Background] El-Shehaby A, Darweesh H, El-Khatib M, Momtaz M, Marzouk S, El-Shaarawy N, Emad Y. Correlations of urinary biomarkers, TNF-like weak inducer of apoptosis (TWEAK), osteoprotegerin (OPG), monocyte chemoattractant protein-1 (MCP-1), and IL-8 with lupus nephritis. J Clin Immunol. 2011 Oct;31(5):848-56. doi: 10.1007/s10875-011-9555-1. Epub 2011 Jun 21. PMID 21691937
- [Background] Wada T, Furuichi K, Sakai N, Iwata Y, Yoshimoto K, Shimizu M, Takeda SI, Takasawa K, Yoshimura M, Kida H, Kobayashi KI, Mukaida N, Naito T, Matsushima K, Yokoyama H. Up-regulation of monocyte chemoattractant protein-1 in tubulointerstitial lesions of human diabetic nephropathy. Kidney Int. 2000 Oct;58(4):1492-9. doi: 10.1046/j.1523-1755.2000.00311.x. PMID 11012884
- [Background] Ommen SR, Nishimura RA, Appleton CP, Miller FA, Oh JK, Redfield MM, Tajik AJ. Clinical utility of Doppler echocardiography and tissue Doppler imaging in the estimation of left ventricular filling pressures: A comparative simultaneous Doppler-catheterization study. Circulation. 2000 Oct 10;102(15):1788-94. doi: 10.1161/01.cir.102.15.1788. PMID 11023933
- [Background] Redfield MM, Jacobsen SJ, Burnett JC Jr, Mahoney DW, Bailey KR, Rodeheffer RJ. Burden of systolic and diastolic ventricular dysfunction in the community: appreciating the scope of the heart failure epidemic. JAMA. 2003 Jan 8;289(2):194-202. doi: 10.1001/jama.289.2.194. PMID 12517230
- [Background] Kuznetsova T, Herbots L, Lopez B, Jin Y, Richart T, Thijs L, Gonzalez A, Herregods MC, Fagard RH, Diez J, Staessen JA. Prevalence of left ventricular diastolic dysfunction in a general population. Circ Heart Fail. 2009 Mar;2(2):105-12. doi: 10.1161/CIRCHEARTFAILURE.108.822627. Epub 2009 Feb 10. PMID 19808325
- [Background] Samdarshi TE, Taylor HA, Edwards DQ, Liebson PR, Sarpong DF, Shreenivas SS, Howard G, Garrison RJ, Fox ER. Distribution and determinants of Doppler-derived diastolic flow indices in African Americans: the Jackson Heart Study (JHS). Am Heart J. 2009 Aug;158(2):209-16. doi: 10.1016/j.ahj.2009.05.020. PMID 19619696
- [Background] Sattar N. Inflammation and endothelial dysfunction: intimate companions in the pathogenesis of vascular disease? Clin Sci (Lond). 2004 May;106(5):443-5. doi: 10.1042/CS20040019. PMID 14741042
- [Background] Taubes G. Cardiovascular disease. Does inflammation cut to the heart of the matter? Science. 2002 Apr 12;296(5566):242-5. doi: 10.1126/science.296.5566.242. No abstract available. PMID 11951014
- [Background] Schwartz CJ, Valente AJ, Sprague EA, Kelley JL, Nerem RM. The pathogenesis of atherosclerosis: an overview. Clin Cardiol. 1991 Feb;14(2 Suppl 1):I1-16. doi: 10.1002/clc.4960141302. PMID 2044253
- [Background] Peters A, Frohlich M, Doring A, Immervoll T, Wichmann HE, Hutchinson WL, Pepys MB, Koenig W. Particulate air pollution is associated with an acute phase response in men; results from the MONICA-Augsburg Study. Eur Heart J. 2001 Jul;22(14):1198-204. doi: 10.1053/euhj.2000.2483. PMID 11440492
- [Background] Kaufmann BA, Carr CL, Belcik JT, Xie A, Yue Q, Chadderdon S, Caplan ES, Khangura J, Bullens S, Bunting S, Lindner JR. Molecular imaging of the initial inflammatory response in atherosclerosis: implications for early detection of disease. Arterioscler Thromb Vasc Biol. 2010 Jan;30(1):54-9. doi: 10.1161/ATVBAHA.109.196386. Epub 2009 Oct 15. PMID 19834105
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Matsushita K, Mahmoodi BK, Woodward M, Emberson JR, Jafar TH, Jee SH, Polkinghorne KR, Shankar A, Smith DH, Tonelli M, Warnock DG, Wen CP, Coresh J, Gansevoort RT, Hemmelgarn BR, Levey AS; Chronic Kidney Disease Prognosis Consortium. Comparison of risk prediction using the CKD-EPI equation and the MDRD study equation for estimated glomerular filtration rate. JAMA. 2012 May 9;307(18):1941-51. doi: 10.1001/jama.2012.3954. PMID 22570462
- [Background] Woodward M. Epidemiology: Study Design and Data Analysis. Third ed. CRC Press; 2014.
- [Background] Devereux RB, Alonso DR, Lutas EM, Gottlieb GJ, Campo E, Sachs I, Reichek N. Echocardiographic assessment of left ventricular hypertrophy: comparison to necropsy findings. Am J Cardiol. 1986 Feb 15;57(6):450-8. doi: 10.1016/0002-9149(86)90771-x. PMID 2936235
- [Background] Nadkarni GN BE. Apolipoprotein L1 Gene Variants Associate with Increased Systolic and Diastolic Blood Pressure in Younger African Americans Independent of Renal Function American Society of Nephrology Kidney Week. Atlanta, GA2013.
- [Background] Mo VY, De Lemos JA. Individualizing therapy in acute coronary syndromes: using a multiple biomarker approach for diagnosis, risk stratification, and guidance of therapy. Curr Cardiol Rep. 2004 Jul;6(4):273-8. doi: 10.1007/s11886-004-0076-x. PMID 15182604
- [Background] Morrow DA, Braunwald E. Future of biomarkers in acute coronary syndromes: moving toward a multimarker strategy. Circulation. 2003 Jul 22;108(3):250-2. doi: 10.1161/01.CIR.0000078080.37974.D2. No abstract available. PMID 12876133
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Quyyumi AA. Circulating endothelial progenitor cells as novel biological determinants of vascular function and risk. Can J Cardiol. 2004 Aug;20 Suppl B:44B-48B. PMID 15309205
- [Background] Ridker PM. Role of inflammatory biomarkers in prediction of coronary heart disease. Lancet. 2001 Sep 22;358(9286):946-8. doi: 10.1016/S0140-6736(01)06112-8. No abstract available. PMID 11583743
- [Background] Pearson TA, Mensah GA, Alexander RW, Anderson JL, Cannon RO 3rd, Criqui M, Fadl YY, Fortmann SP, Hong Y, Myers GL, Rifai N, Smith SC Jr, Taubert K, Tracy RP, Vinicor F; Centers for Disease Control and Prevention; American Heart Association. Markers of inflammation and cardiovascular disease: application to clinical and public health practice: A statement for healthcare professionals from the Centers for Disease Control and Prevention and the American Heart Association. Circulation. 2003 Jan 28;107(3):499-511. doi: 10.1161/01.cir.0000052939.59093.45. No abstract available. PMID 12551878
- [Background] deFilippi CR, de Lemos JA, Christenson RH, Gottdiener JS, Kop WJ, Zhan M, Seliger SL. Association of serial measures of cardiac troponin T using a sensitive assay with incident heart failure and cardiovascular mortality in older adults. JAMA. 2010 Dec 8;304(22):2494-502. doi: 10.1001/jama.2010.1708. Epub 2010 Nov 15. PMID 21078811
- [Background] de Lemos JA, Drazner MH, Omland T, Ayers CR, Khera A, Rohatgi A, Hashim I, Berry JD, Das SR, Morrow DA, McGuire DK. Association of troponin T detected with a highly sensitive assay and cardiac structure and mortality risk in the general population. JAMA. 2010 Dec 8;304(22):2503-12. doi: 10.1001/jama.2010.1768. PMID 21139111
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Nohria A, Gerhard-Herman M, Creager MA, Hurley S, Mitra D, Ganz P. Role of nitric oxide in the regulation of digital pulse volume amplitude in humans. J Appl Physiol (1985). 2006 Aug;101(2):545-8. doi: 10.1152/japplphysiol.01285.2005. Epub 2006 Apr 13. PMID 16614356
- [Background] Sawit S MM, Garcia-Alvarez A, Fahima DK, Maceda C, Moline J. Evidence of Impaired Vascular Reactivity Following Dust Exposure in Participants of the World Trade Center Medical Monitoring and Treatment Program. New York City: Mount Sinai School of Medicine; 2011.